CLINICAL TRIAL: NCT02202434
Title: REPRISE III: Repositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of Lotus™ Valve System - Randomized Clinical Evaluation
Brief Title: Safety and Efficacy Study of Lotus Valve for Transcatheter Aortic Valve Replacement
Acronym: REPRISE III
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: RCT/Roll-in completed. CAS/21mm/Nested Registry terminated (investigational device is no longer available)
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2282
Record Dates: First submitted 2014-07-21; First posted 2014-07-29 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Lotus Valve System - Randomized (Experimental): Transcatheter aortic valve replacement (TAVR) with Lotus Valve System
  Interventions: Device: Lotus Valve System
- CoreValve TAVR System - Randomized (Active Comparator): Transcatheter aortic valve replacement (TAVR) with CoreValve/Evolut R Transcatheter Aortic Valve Replacement System
  Interventions: Device: CoreValve/Evolut R Transcatheter Aortic Valve Replacement System
- Lotus Valve Sytem - Single-arm 21mm Cohort (Experimental): Transcatheter aortic valve replacement (TAVR) with 21mm Lotus Valve System
  Interventions: Device: Lotus Valve System
- Lotus Valve System - Single-arm Continued Access Cohort (Experimental): Transcatheter aortic valve replacement (TAVR) with Lotus Valve System
  Interventions: Device: Lotus Valve System
- Lotus Valve System - Single-arm Roll-in Cohort (Experimental): Transcatheter aortic valve replacement (TAVR) with Lotus Valve System
  Interventions: Device: Lotus Valve System
- LOTUS Edge Valve System - Single-arm Edge Nested Registry (Experimental): Transcatheter aortic valve replacement (TAVR) with 23mm, 25mm and 27mm LOTUS Edge Valve System.
  Interventions: Device: LOTUS Edge Valve System

INTERVENTIONS:
Device: Lotus Valve System — Procedure: Transcatheter aortic valve replacement (TAVR)
  Arms: Lotus Valve System - Randomized; Lotus Valve System - Single-arm Continued Access Cohort; Lotus Valve System - Single-arm Roll-in Cohort; Lotus Valve Sytem - Single-arm 21mm Cohort
Device: CoreValve/Evolut R Transcatheter Aortic Valve Replacement System — Procedure: Transcatheter aortic valve replacement (TAVR)
  Arms: CoreValve TAVR System - Randomized
Device: LOTUS Edge Valve System — Procedure: Transcatheter aortic valve replacement (TAVR)
  Arms: LOTUS Edge Valve System - Single-arm Edge Nested Registry

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Lotus™ Valve System and LOTUS Edge™ Valve System for transcatheter aortic valve replacement (TAVR) in symptomatic subjects with calcific, severe native aortic stenosis who are considered at extreme or high risk for surgical valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has documented calcific, severe native aortic stenosis with an initial aortic valve area (AVA) of ≤1.0 cm2 (or AVA index of ≤0.6 cm2/m2) and a mean pressure gradient >40 mm Hg or jet velocity >4.0 m/s, as measured by echocardiography and/or invasive hemodynamics
2. Subject has a documented aortic annulus size of ≥18 mm and ≤29 mm based on the center's assessment of pre-procedure diagnostic imaging (and confirmed by the Case Review Committee [CRC]) and, for the randomized cohort, is deemed treatable with an available size of both test and control device. For the U.S. Continued Access Study cohort the acceptable aortic annulus size is ≥20 mm and ≤27 mm.
3. Subject has symptomatic aortic valve stenosis with New York Heart Association (NYHA) Functional Class ≥ II
4. There is agreement by the heart team (which must include a site investigator interventionalist and a site investigator cardiac surgeon) that subject is at high or extreme operative risk for surgical valve replacement (see note below for definitions of extreme and high risk, the required level of surgical assessment, and CRC confirmation) and that TAVR is appropriate. Additionally, subject has at least one of the following.

   * Society of Thoracic Surgeons (STS) score ≥8% -OR-
   * If STS <8, subject has at least one of the following conditions: Hostile chest, porcelain aorta, severe pulmonary hypertension (>60 mmHg), prior chest radiation therapy, coronary artery bypass graft(s) at risk with re-operation, severe lung disease (need for supplemental oxygen, forced expiratory volume in 1 second [FEV1] <50% of predicted, diffusing capacity of the lungs for carbon monoxide [DLCO] <60%, or other evidence of severe pulmonary dysfunction), neuromuscular disease that creates risk for mechanical ventilation or rehabilitation after surgical aortic valve replacement, orthopedic disease that creates risk for rehabilitation after surgical aortic valve replacement, Childs Class A or B liver disease (subjects with Childs Class C disease are not eligible for inclusion in this trial), frailty as indicated by at least one of the following: 5-meter walk >6 seconds, Katz Assessment of Daily Living (Katz ADL) score of 3/6 or less, body mass index <21, wheelchair bound, unable to live independently, age ≥90 years, other evidence that subject is at high or extreme risk for surgical valve replacement (CRC must confirm agreement with site heart team that subject meets high or extreme risk definition)
5. Heart team (which must include a cardiac interventionalist and an experienced cardiac surgeon) assessment that the subject is likely to benefit from valve replacement.
6. Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent.
7. Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.

Note: Extreme operative risk and high operative risk are defined as follows: Extreme Operative Risk: Predicted operative mortality or serious, irreversible morbidity risk ≥50% at 30 days; High Operative Risk: Predicted operative mortality or serious, irreversible morbidity risk ≥15% at 30 days. Risk of operative mortality and morbidity must be assessed via an in-person evaluation by a center cardiac surgeon and must be confirmed by the CRC (which must include an experienced cardiac surgeon).

Exclusion Criteria:

1. Subject has a congenital unicuspid or bicuspid aortic valve.
2. Subject has had an acute myocardial infarction (MI) within 30 days prior to the index procedure (defined as Q-wave MI or non-Q-wave MI with total creatine kinase (CK) elevation ≥ twice normal in the presence of creatine kinase-myoglobin band (CK-MB) elevation and/or troponin elevation).
3. Subject has had a cerebrovascular accident or transient ischemic attack within the past 6 months prior to study enrollment.
4. Subject has end-stage renal disease or has glomerular filtration rate (GFR) <20 (based on Cockcroft-Gault formula).
5. Subject has a pre-existing prosthetic aortic or mitral valve.
6. Subject has severe (4+) aortic, tricuspid, or mitral regurgitation.
7. Subject has a need for emergency surgery for any reason.
8. Subject has a history of endocarditis within 6 months of index procedure or evidence of an active systemic infection or sepsis.
9. Subject has echocardiographic evidence of new intra-cardiac mass, vegetation or intraventricular or paravalvular thrombus requiring intervention.
10. Subject has (hemoglobin) Hgb <9 g/dL, platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.
11. Subject requires chronic anticoagulation therapy after the implant procedure and cannot be treated with warfarin (other anticoagulants are not permitted in the first month) for at least 1 month concomitant with either aspirin or clopidogrel.
12. Subject has had a gastrointestinal bleed requiring hospitalization or transfusion within the past 3 months, or has other clinically significant bleeding diathesis or coagulopathy that would preclude treatment with required antiplatelet regimen, or will refuse transfusions.
13. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all P2Y12 inhibitors, heparin, nickel, tantalum, titanium, or polyurethanes.
14. Subject has a life expectancy of less than 12 months due to non-cardiac, comorbid conditions based on the assessment of the investigator at the time of enrollment.
15. Subject has hypertrophic obstructive cardiomyopathy.
16. Subject has any therapeutic invasive cardiac or vascular procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty or pacemaker implantation, which are allowed).
17. Subject has untreated coronary artery disease, which in the opinion of the treating physician is clinically significant and requires revascularization.
18. Subject has severe left ventricular dysfunction with ejection fraction <20%.
19. Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
20. Subject has severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely, marked tortuosity, significant narrowing of the abdominal aorta, severe unfolding of the thoracic aorta, or symptomatic carotid or vertebral disease).
21. Subject has thick (>5 mm) protruding or ulcerated atheroma in the aortic arch
22. Subject has arterial access that is not acceptable for the test and control device delivery systems as defined in the device Instructions For Use.
23. Subject has current problems with substance abuse (e.g., alcohol, etc.).
24. Subject is participating in another investigational drug or device study that has not reached its primary endpoint.
25. Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation. Enrollment is permissible after permanent pacemaker implantation.
26. Subject has severe incapacitating dementia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1425 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizik, MD, Principal Investigator — Scottsdale Healthcare - Shea; Michael J Reardon, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (58):
- United States (49):
  - Banner Good Samaritan, Phoenix, Arizona
  - Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Scripps Clinic, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Veteran's Administration Palo Alto Medical Center, Palo Alto, California
  - University of California at Davis Medical Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Mease Healthcare System, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - University of Miami Hospital, Miami, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Evanston Hospital, Evanston, Illinois
  - St. John's Hospital - Prairie Cardiovascular Consultants, Springfield, Illinois
  - St. Vincent's Hospital, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - Union Memorial Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cardiac & Vascular Rearch Center of Northern Michigan - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Abbott Northwestern Hospital - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine - Barnes Jewish Medical Center, St Louis, Missouri
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Kaleida Health, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - NC Heart and Vascular Research - Rex Hospital, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Ohio Health Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - Methodist Heart Hospital, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (2):
  - The Prince Charles Hospital, Chermside, Queensland
  - Monash Medical Centre, Clayton, Victoria
- Canada (2):
  - Providence Health - St. Paul's Hospital, Vancouver, British Columbia
  - McGill University Health Centre, Royal Victoria Hospital, Montreal, Quebec
- France (2):
  - Clinique Pasteur, Toulouse, Midi-Pyrenees
  - Centre Hôpital Universitaire Rangueil, Toulouse
- Germany (2):
  - Herzzentrum Universität Leipzig, Leipzig, Saxony
  - Universitares Herzzentrum UKE (Hamburg), Hamburg
- Erasmus MC - University Medical Center Rotterdam, Rotterdam, Netherlands

REFERENCES:
- [Derived] Rizik DG, Rajagopal V, Makkar RR, Bajwa T, Kleiman NS, Linke A, Kereiakes DJ, Waksman R, Thourani VH, Stoler RC, Mishkel GJ, Iyer VS, Buchbinder M, Gotberg M, Bjursten H, Allocco DJ, Reardon MJ. Long-term Outcomes of Transcatheter Aortic Valve Replacement With the Lotus Valve vs CoreValve/EvolutR: A Secondary Analysis of the REPRISE III Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2238792. doi: 10.1001/jamanetworkopen.2022.38792. PMID 36301543
- [Derived] Goel K, O'Leary JM, Barker CM, Levack M, Rajagopal V, Makkar RR, Bajwa T, Kleiman N, Linke A, Kereiakes DJ, Waksman R, Allocco DJ, Rizik DG, Reardon MJ, Lindman BR. Clinical Implications of Physical Function and Resilience in Patients Undergoing Transcatheter Aortic Valve Replacement. J Am Heart Assoc. 2020 Sep;9(17):e017075. doi: 10.1161/JAHA.120.017075. Epub 2020 Aug 28. PMID 32856530
- [Derived] Meduri CU, Kereiakes DJ, Rajagopal V, Makkar RR, O'Hair D, Linke A, Waksman R, Babliaros V, Stoler RC, Mishkel GJ, Rizik DG, Iyer VS, Schindler J, Allocco DJ, Meredith IT, Feldman TE, Reardon MJ. Pacemaker Implantation and Dependency After Transcatheter Aortic Valve Replacement in the REPRISE III Trial. J Am Heart Assoc. 2019 Nov 5;8(21):e012594. doi: 10.1161/JAHA.119.012594. Epub 2019 Oct 23. PMID 31640455
- [Derived] Reardon MJ, Feldman TE, Meduri CU, Makkar RR, O'Hair D, Linke A, Kereiakes DJ, Waksman R, Babliaros V, Stoler RC, Mishkel GJ, Rizik DG, Iyer VS, Gleason TG, Tchetche D, Rovin JD, Lhermusier T, Carrie D, Hodson RW, Allocco DJ, Meredith IT; Reprise III Investigators. Two-Year Outcomes After Transcatheter Aortic Valve Replacement With Mechanical vs Self-expanding Valves: The REPRISE III Randomized Clinical Trial. JAMA Cardiol. 2019 Mar 1;4(3):223-229. doi: 10.1001/jamacardio.2019.0091. PMID 30810703
- [Derived] Asch FM, Vannan MA, Singh S, Khandheria B, Little SH, Allocco DJ, Meredith IT, Feldman TE, Reardon MJ, Weissman NJ. Hemodynamic and Echocardiographic Comparison of the Lotus and CoreValve Transcatheter Aortic Valves in Patients With High and Extreme Surgical Risk: An Analysis From the REPRISE III Randomized Controlled Trial. Circulation. 2018 Jun 12;137(24):2557-2567. doi: 10.1161/CIRCULATIONAHA.118.034129. Epub 2018 Mar 12. PMID 29530883
- [Derived] Feldman TE, Reardon MJ, Rajagopal V, Makkar RR, Bajwa TK, Kleiman NS, Linke A, Kereiakes DJ, Waksman R, Thourani VH, Stoler RC, Mishkel GJ, Rizik DG, Iyer VS, Gleason TG, Tchetche D, Rovin JD, Buchbinder M, Meredith IT, Gotberg M, Bjursten H, Meduri C, Salinger MH, Allocco DJ, Dawkins KD. Effect of Mechanically Expanded vs Self-Expanding Transcatheter Aortic Valve Replacement on Mortality and Major Adverse Clinical Events in High-Risk Patients With Aortic Stenosis: The REPRISE III Randomized Clinical Trial. JAMA. 2018 Jan 2;319(1):27-37. doi: 10.1001/jama.2017.19132. PMID 29297076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 912 subjects randomized from 22Sep2014 to 24Dec2015. 102 subjects enrolled in the Roll-in cohort. 295 subjects enrolled in the US CAS from 25Feb2016 to 23Feb2017. Enrollment in the LOTUS Edge Valve System - Single-arm Edge Nested Reg is ongoing.
  Enrollment in the LOTUS Edge Valve System - Single-arm 29mm Reg and Roll-in Cohorts has not begun.
Pre-assignment Details: The non-randomized Roll-In phase with only the test device was for centers with no previous experience implanting the Lotus Valve System. Each performed at least two Roll-In cases before starting RCT.
  Only cohorts that have completed enrollment, reached primary endpoint and were submitted for regulatory approval are included in the Results Section
Groups:
- CoreValve TAVR System - Randomized: Transcatheter aortic valve replacement (TAVR) with CoreValve Transcatheter Aortic Valve Replacement System
  CoreValve Transcatheter Aortic Valve Replacement System: Procedure: Transcatheter aortic valve replacement (TAVR)
Period: Overall Study
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Started | 607 | 305 | 102 | 295
Completed | 498 | 236 | 87 | 258
Not Completed | 109 | 69 | 15 | 37
Not completed — Death | 70 | 39 | 13 | 27
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Physician Decision | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 14 | 1 | 4
Not completed — Completed Study | 1 | 0 | 0 | 0
Not completed — Visit Missed | 21 | 12 | 0 | 5
Not completed — Other | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data are reported separately for each cohort as pooled mean and standard deviations across cohorts do not provide meaningful data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort | Total
Number analyzed (Participants) | 607 | 305 | 102 | 295 | 1309
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Lotus Valve System - Randomized | 82.8 (7.1) | 0 (0) | 0 (0) | 0 (0) | 82.8 (7.1)
  CoreValve TAVR System - Randomize | 0 (0) | 82.9 (7.6) | 0 (0) | 0 (0) | 82.9 (7.6)
  Lotus Valve System - Single-arm Roll-in Cohort | 0 (0) | 0 (0) | 83.6 (6.9) | 0 (0) | 83.6 (6.9)
  Lotus Valve System - Single-arm Continued Access | 0 (0) | 0 (0) | 0 (0) | 81.7 (6.6) | 81.7 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 159 | 52 | 137 | 652
  Male | 303 | 146 | 50 | 158 | 657
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Subjects were allowed to select more than one option.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1 | 1 | 3
    Asian | 3 | 2 | 0 | 4 | 9
    Black, of African Heritage | 17 | 11 | 4 | 13 | 45
    Caucasian | 537 | 271 | 93 | 271 | 1172
    Hispanic or Latino | 18 | 2 | 4 | 6 | 30
    Native Hawaiian or other Pacific Islander | 2 | 1 | 0 | 0 | 3
    Other | 3 | 4 | 0 | 1 | 8
    Unknown or Not Reported | 28 | 14 | 1 | 0 | 43
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 2 | 0 | 4
  Netherlands | 4 | 2 | 0 | 0 | 6
  United States | 531 | 261 | 100 | 295 | 1187
  Australia | 15 | 8 | 0 | 0 | 23
  France | 23 | 13 | 0 | 0 | 36
  Germany | 33 | 20 | 0 | 0 | 53
Society of Thoracic Surgeons (STS) Risk Score [Mean (Standard Deviation); unit: Percent] — The Society of Thoracic Surgeons Score is a risk model used to predict a subject's risk of mortality and morbidities for the most commonly performed cardiac surgeries. The model is a percentage score from 0 to 100 where a lower score means a lower risk and higher score means a higher risk.
  Percent
    Lotus Valve System - Randomized | 6.7 (4.0) | 0 (0) | 0 (0) | 0 (0) | 6.7 (4.0)
    CoreValve TAVR System - Randomized | 0 (0) | 6.9 (4.1) | 0 (0) | 0 (0) | 6.9 (4.1)
    Lotus Valve System - Single-arm Roll-in Cohort | 0 (0) | 0 (0) | 7.0 (4.9) | 0 (0) | 7.0 (4.9)
    Lotus Valve System - Single-arm Continued Access | 0 (0) | 0 (0) | 0 (0) | 5.4 (2.9) | 5.4 (2.9)
European System for Cardiac Operative Risk Evaluation (EuroSCORE) [Mean (Standard Deviation); unit: Percent] — The European System for Cardiac Operative Risk Evaluation is a risk model where if a risk factor is present in a subject, a weight or number is assigned. The weights are added to give an approximate percent predicted mortality. A higher score means a higher risk and a lower score means a lower risk.
  Percent
    Lotus Valve System - Randomized | 6.4 (5.5) | 0 (0) | 0 (0) | 0 (0) | 6.4 (5.5)
    CoreValve TAVR System - Randomized | 0 (0) | 6.4 (5.5) | 0 (0) | 0 (0) | 6.4 (5.5)
    Lotus Valve System - Single-arm Roll-in Cohort | 0 (0) | 0 (0) | 6.4 (6.5) | 0 (0) | 6.4 (6.5)
    Lotus Valve System - Single-arm Continued Access | 0 (0) | 0 (0) | 0 (0) | 5.3 (5.9) | 5.3 (5.9)
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — New York Heart Association Classification is a system for defining cardiac disease and related functional limitations into four broad categorizations. The categories range from NYHA I (No limitations) to NYHA IV (inability to carry out any physical activity without discomfort).
  Participants
    NYHA I | 0 | 0 | 0 | 0 | 0
    NYHA II | 174 | 98 | 22 | 108 | 402
    NYHA III | 386 | 186 | 70 | 171 | 813
    NYHA IV | 47 | 21 | 10 | 16 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Events Included in the Primary Safety Endpoint
Description: Composite of all-cause mortality, stroke, life-threatening and major bleeding events, stage 2 or 3 acute kidney injury, or major vascular complications
Time Frame: 30 days following procedure
Population: Implanted population - all subjects who sign an Informed Consent Form, are enrolled in the trial, and are implanted with the assigned, randomized study device. The Primary and Secondary Endpoints (Outcome Measures 1-3) are only applicable to the two Randomized arms of the study.
Measure: Number; unit: Percent of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized
Number analyzed (Participants) | 577 | 297
Percent of participants | 20.3 | 17.2
Statistical Analysis 1: Comparison: Lotus Valve System - Randomized vs CoreValve TAVR System - Randomized; Test type: Non-Inferiority — 10.5% non-inferiority margin; p = 0.0027, Farrington-Manning; Difference in Percentages = 3.1, 97.5% CI 1-sided [upper limit 8.32]

2. Primary Outcome: Percentage of Participants With Events Included in the Primary Effectiveness Endpoint
Description: Composite of all-cause mortality, disabling stroke, or moderate or greater paravalvular aortic regurgitation (based on core lab assessment).
Time Frame: 1 year following procedure
Population: Non-inferiority analysis - Implanted population - all subjects who sign an Informed Consent Form, are enrolled in the trial, and are implanted with the assigned, randomized study device.
  Superiority analysis - Intent to Treat Population The Primary and Secondary Endpoints (Outcome Measures 1-3) are only applicable to the two Randomized arms.
Measure: Number; unit: Percent of Participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized
Number analyzed (Participants) | 607 | 305
Percent of Participants
  Implanted: number analyzed (Participants) | 577 | 297
  Implanted | 15.4 | 25.5
  Intent to Treat | 15.8 | 26.0
Statistical Analysis 1: Comparison: Lotus Valve System - Randomized vs CoreValve TAVR System - Randomized; Test type: Non-Inferiority — 9.5% Non-Inferiority margin; p < 0.0001, Farrington-Manning; Difference in Percentages = -10.1, 97.5% CI 1-sided [upper limit -4.41]
Statistical Analysis 2: Comparison: Lotus Valve System - Randomized vs CoreValve TAVR System - Randomized; Superiority analysis was only to be run if the non-inferiority analysis was met. Superiority analysis was run on Intent to Treat Population; Test type: Superiority; p = 0.0006, Chi-squared; Difference in Percentages = -10.2, 95% CI 2-sided [-16.3 to -4.0]

3. Secondary Outcome: Percentage of Participants With Moderate or Greater Paravalvular Aortic Regurgitation
Description: Moderate or greater paravalvular aortic regurgitation based on Independent echocardiographic core lab assessment performed using the Unifying 5-Class Grading Scheme for Aortic Regurgitation by Pibarot et al (J Am Coll Cardiol Img 2015: 8: 340-60). The grading scheme ranges from Trace (the least clinically significant) to severe (the most clinically significant).
Time Frame: 1 year following procedure
Population: ITT - all subjects who sign an Informed Consent Form, are enrolled in the trial, and are randomized, whether or not an assigned study device is implanted.
  The Primary and Secondary Endpoints (Outcome Measures 1-3) are only applicable to the two Randomized arms of the study.
Measure: Number; unit: Percent of Participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized
Number analyzed (Participants) | 607 | 305
Percent of Participants | 0.9 | 6.9
Statistical Analysis 1: Comparison: Lotus Valve System - Randomized vs CoreValve TAVR System - Randomized; Test type: Superiority; p < 0.0001, Chi-squared; Difference in Percentages = -6.1, 95% CI 2-sided [-9.6 to -2.6]

4. Other Pre Specified Outcome: Percentage of Participants With Successful Deployment of the Study Valve
Description: Successful deployment of the study valve
Time Frame: at discharge or 7 days post-procedure (whichever comes first)
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants | 97.8 | 99.0 | 99.0 | 96.6

5. Other Pre Specified Outcome: Percentage of Participants With Successful Retrieval of the Study Valve if Retrieval is Attempted
Description: Successful retrieval of the study valve if retrieval is attempted
Time Frame: at discharge or 7 days post-procedure (whichever comes first)
Population: Number of Intent to Treat participants who had Retrieval attempted
Measure: Number; unit: Percentage of Participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 40 | 14 | 5 | 24
Percentage of Participants | 100 | 92.9 | 100 | 100

6. Other Pre Specified Outcome: Percentage of Participants With Successful Repositioning of the Study Valve if Repositioning is Attempted
Description: Successful repositioning of the study valve if repositioning is attempted
Time Frame: at discharge or 7 days post-procedure (whichever comes first)
Population: Number of Intent to Treat participants who had Repositioning attempted
Measure: Number; unit: Percentage of Participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 197 | 35 | 46 | 140
Percentage of Participants | 100 | 100 | 100 | 97.1

7. Other Pre Specified Outcome: Percentage of Participants With Each Grade of Aortic Valve Regurgitation in Each Location: Paravalvular, Central, and Combined
Description: Grade of aortic valve regurgitation: paravalvular, central, and combined. An Independent echocardiographic core lab assessment was performed using the Unifying 5-Class Grading Scheme for Aortic Regurgitation for the locations paravalvular, central and combined.
  The grading scheme has a range from Trace to Severe. A grade of Trace is the least clinically significant (better outcome) and a grade of Severe is the most clinically significant (worse outcome).
Time Frame: at discharge or 7 days post-procedure (whichever comes first)
Population: Intent to Treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of Participants
  Central - Trace or Greater | 15.2 | 8.7 | 15.8 | 15.3
  Central - None | 84.8 | 91.3 | 84.2 | 84.7
  Central - Trace/Trivial | 6.1 | 1.8 | 6.3 | 4.0
  Central - Mild | 4.2 | 0.7 | 3.2 | 4.7
  Central - Mild-Moderate | 0.0 | 0.0 | 0.0 | 0.0
  Central - Moderate | 0.0 | 0.4 | 1.1 | 0.0
  Central - Moderate-Severe | 0.0 | 0.0 | 0.0 | 0.0
  Central - Severe | 0.0 | 0.0 | 0.0 | 0.0
  Central - Moderate or Greater | 0.0 | 0.4 | 1.1 | 0.0
  Central - AR but Severity Not Evaluable | 4.9 | 5.8 | 5.3 | 6.6
  Paravalvular - Trace or Greater | 26.9 | 72.6 | 28.4 | 28.5
  Paravalvular - None | 73.1 | 27.4 | 71.6 | 71.5
  Paravalvular - Trace/Trivial | 10.5 | 18.1 | 12.6 | 2.9
  Paravalvular - Mild | 11.8 | 46.9 | 12.6 | 18.2
  Paravalvular - Mild-Moderate | 0.0 | 0.0 | 0.0 | 0.0
  Paravalvular - Moderate | 0.4 | 3.6 | 0.0 | 0.4
  Paravalvular - Moderate-Severe | 0.0 | 0.0 | 0.0 | 0.0
  Paravalvular - Severe | 0.0 | 0.0 | 0.0 | 0.0
  Paravalvular - Moderate or Greater | 0.4 | 3.6 | 0.0 | 0.4
  Paravalvular - AR but Severity Not Evaluable | 4.3 | 4.0 | 3.2 | 6.9
  Total - Trace or Greater | 35.1 | 73.3 | 36.8 | 34.7
  Total - None | 64.9 | 26.7 | 63.2 | 65.3
  Total - Trace/Trivial | 17.4 | 18.4 | 20.0 | 8.8
  Total - Mild | 15.4 | 48.7 | 15.8 | 24.5
  Total - Mild-Moderate | 0.0 | 0.0 | 0.0 | 0.0
  Total - Moderate | 0.9 | 4.3 | 1.1 | 0.4
  Total - Moderate-Severe | 0.0 | 0.0 | 0.0 | 0.0
  Total - Severe | 0.0 | 0.0 | 0.0 | 0.0
  Total - Moderate or Greater | 0.9 | 4.3 | 1.1 | 0.4
  Total - AR but Severity Not Evaluable | 1.4 | 1.8 | 0.0 | 1.1

8. Other Pre Specified Outcome: Percentage of Participants With Clinical Procedural Success
Description: Defined as implantation of the study device in the absence of death, disabling stroke, major vascular complications, and life-threatening or major bleeding
Time Frame: 30 days post procedure
Population: Intent to Treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of Participants | 81.4 | 84.6 | 81.4 | 81.0

9. Other Pre Specified Outcome: Percentage of Participants With Procedural Success
Description: Defined as absence of procedural mortality, correct positioning of a single transcatheter valve into the proper anatomical location , intended performance of the study device (effective orifice area [EOA] >0.9 cm2 for body surface area (BSA) <1.6 m2 and EOA >1.1 cm2 for BSA ≥1.6 m2 plus either a mean aortic valve gradient <20 mm Hg or a peak velocity <3m/sec, and no moderate or severe prosthetic valve aortic regurgitation) plus no serious adverse events
Time Frame: 30 days post procedure
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants | 32.0 | 39.2 | 33.3 | 29.3

10. Other Pre Specified Outcome: Additional Indications of Prosthetic Aortic Valve Performance as Measured by Transthoracic Echocardiography 1
Description: Assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, and peak aortic velocity
Time Frame: assessed at discharge, 30 days, 6 months, and 1, 2, 3, 4, and 5 years post index procedure, at discharge, 30 days, 6 months, and 1 year post index procedure reported.
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
cm^2
  Discharge or 7 Days - Aortic Valve Area | 1.65 (0.47) | 1.96 (0.52) | 1.70 (0.49) | 1.61 (0.42)
  30 Days - Aortic Valve Area | 1.59 (0.45) | 1.98 (0.51) | 1.62 (0.46) | 1.55 (0.41)
  6 Months - Aortic Valve Area | 1.46 (0.46) | 1.74 (0.55) | 1.55 (0.45) | 1.56 (0.47)
  1 Year - Aortic Valve Area | 1.49 (0.45) | 1.69 (0.52) | 1.53 (0.49) | 1.51 (0.46)

11. Other Pre Specified Outcome: Additional Indications of Prosthetic Aortic Valve Performance as Measured by Transthoracic Echocardiography 2
Description: Assessed by an independent core laboratory - mean and peak aortic gradients
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
mmHg
  Discharge or 7 Days - Mean Aortic Valve Gradient | 12.20 (5.21) | 8.19 (3.98) | 12.13 (5.13) | 12.50 (6.01)
  Discharge or 7 Days - Peak Aortic Gradient | 22.28 (10.23) | 15.21 (7.20) | 21.58 (8.55) | 22.89 (10.91)
  30 Days - Mean Aortic Valve Gradient | 12.00 (6.08) | 7.25 (3.44) | 12.76 (8.24) | 12.24 (6.73)
  30 Days - Peak Aortic Gradient | 21.46 (10.27) | 13.59 (6.21) | 23.02 (13.43) | 22.56 (11.44)
  6 Months - Mean Aortic Valve Gradient | 11.93 (5.21) | 7.89 (4.24) | 12.33 (5.89) | 12.20 (5.42)
  6 Months - Peak Aortic Gradient | 22.24 (9.82) | 14.84 (7.46) | 22.85 (10.60) | 22.68 (9.81)
  1 Year - Mean Aortic Valve Gradient | 12.29 (5.83) | 7.89 (3.48) | 12.30 (7.39) | 12.68 (5.62)
  1 Year - Peak Aortic Gradient | 22.74 (10.53) | 15.22 (6.44) | 22.03 (12.05) | 23.75 (9.83)

12. Other Pre Specified Outcome: Additional Indications of Prosthetic Aortic Valve Performance as Measured by Transthoracic Echocardiography 3
Description: Assessed by an independent core laboratory - peak aortic velocity
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
m/s
  Discharge or 7 Days - Peak Aortic Velocity | 2.30 (0.48) | 1.89 (0.45) | 2.28 (0.44) | 2.33 (0.53)
  30 Days - Peak Aortic Velocity | 2.26 (0.46) | 1.80 (0.40) | 2.33 (0.58) | 2.31 (0.53)
  6 Months - Peak Aortic Velocity | 2.30 (0.46) | 1.87 (0.44) | 2.32 (0.49) | 2.33 (0.49)
  1 Year - Peak Aortic Velocity | 2.33 (0.51) | 1.91 (0.41) | 2.28 (0.55) | 2.39 (0.47)

13. Other Pre Specified Outcome: Percentage of Participants With Additional Indications of Prosthetic Aortic Valve Performance as Measured by Transthoracic Echocardiography 4
Description: as for outcome 7
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge Paravalvular - Trace or Greater | 26.9 | 72.6 | 28.4 | 28.5
  Discharge Paravalvular None | 73.1 | 27.4 | 71.6 | 71.5
  Discharge Paravalvular Trace/Trivial | 10.5 | 18.1 | 12.6 | 2.9
  Discharge Paravalvular Mild | 11.8 | 46.9 | 12.6 | 18.2
  Discharge Paravalvular Mild-Moderate | 0.0 | 0.0 | 0.0 | 0.0
  Discharge Paravalvular Moderate | 0.4 | 3.6 | 0.0 | 0.4
  Discharge Paravalvular Moderate-Severe | 0.0 | 0.0 | 0.0 | 0.0
  Discharge Paravalvular Severe | 0.0 | 0.0 | 0.0 | 0.0
  Discharge Paravalvular Moderate or Greater | 0.4 | 3.6 | 0.0 | 0.4
  Discharge ParavalvularAR but Severity not evaluabl | 4.3 | 4.0 | 3.2 | 6.9
  30 Day Paravalvular - Trace or Greater | 27.5 | 75.5 | 30.0 | 27.3
  30 Day Paravalvular None | 72.5 | 24.5 | 70.0 | 72.7
  30 Day Paravalvular Trace/Trivial | 10.7 | 14.7 | 10.0 | 2.5
  30 Day Paravalvular Mild | 10.7 | 48.7 | 15.0 | 18.5
  30 Day Paravalvular Mild-Moderate | 0.0 | 0.0 | 0.0 | 0.0
  30 Day Paravalvular Moderate | 0.4 | 7.2 | 1.0 | 1.5
  30 Day Paravalvular Moderate-Severe | 0.2 | 0.0 | 0.0 | 0.0
  30 Day Paravalvular Severe | 0.0 | 0.0 | 0.0 | 0.0
  30 Day Paravalvular Moderate or Greater | 0.6 | 7.2 | 1.0 | 1.5
  30 Day Paravalvular AR but Severity not evaluable | 5.5 | 4.9 | 4.0 | 4.7
  6 Month Paravalvular - Trace or Greater | 22.3 | 62.7 | 23.8 | 26.9
  6 Month Paravalvular None | 77.7 | 37.3 | 76.2 | 73.1
  6 Month Paravalvular Trace/Trivial | 4.2 | 6.8 | 7.1 | 4.3
  6 Month Paravalvular Mild | 11.5 | 42.4 | 14.3 | 19.8
  6 Month Paravalvular Mild-Moderate | 0.0 | 0.0 | 0.0 | 0.0
  6 Month Paravalvular Moderate | 0.4 | 4.7 | 0.0 | 0.0
  6 Month Paravalvular Moderate-Severe | 0.2 | 0.0 | 0.0 | 0.0
  6 Month Paravalvular Severe | 0.0 | 0.0 | 0.0 | 0.0
  6 Month Paravalvular Moderate or Greater | 0.6 | 4.7 | 0.0 | 0.0
  6 Month Paravalvular AR but Severity not evaluable | 5.9 | 8.9 | 2.4 | 2.8
  1 Year Paravalvular - Trace or Greater | 20.1 | 63.0 | 24.4 | 20.6
  1 Year Paravalvular None | 79.9 | 37.0 | 75.6 | 79.4
  1 Year Paravalvular Trace/Trivial | 5.7 | 10.5 | 4.7 | 3.3
  1 Year Paravalvular Mild | 11.3 | 38.8 | 14.0 | 12.3
  1 Year Paravalvular Mild-Moderate | 0.0 | 0.0 | 0.0 | 0.0
  1 Year Paravalvular Moderate | 0.9 | 5.9 | 0.0 | 1.2
  1 Year Paravalvular Moderate-Severe | 0.0 | 0.9 | 0.0 | 0.0
  1 Year Paravalvular Severe | 0.0 | 0.0 | 0.0 | 0.0
  1 Year Paravalvular Moderate or Greater | 0.9 | 6.8 | 0.0 | 1.2
  1 Year Paravalvular AR but Severity not evaluable | 2.2 | 6.8 | 5.8 | 3.7

14. Other Pre Specified Outcome: Health Status as Evaluated by Quality of Life Questionnaires
Description: SF-12 and Kansas City Cardiomyopathy - Baseline scores and changes from Baseline at 30 days, 6 months and 1 year
  * SF-12 Item Short Form Health Survey (SF-12): Measures functional health and well-being. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  * Kansas City Cardiomyopathy Questionnaire (KCCQ): Quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life.
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Assessed at Baseline, 1 and 6 months; and 1, 3, and 5 years, at Baseline, 1 and 6 months and 1 Year reported
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Score on a scale
  Baseline SF-12 Physical Summary Score | 31.9 (9.0) | 31.2 (8.9) | 33.8 (10.5) | 32.4 (10.0)
  Baseline SF-12 Mental Health Summary Score | 49.6 (11.6) | 49.0 (11.6) | 49.8 (11.0) | 50.0 (11.4)
  Baseline KC Overall Summary Score | 51.9 (23.5) | 50.7 (22.1) | 52.7 (24.6) | 53.5 (22.8)
  Baseline KC Clinical Summary Score | 55.2 (23.3) | 54.9 (21.9) | 57.3 (23.7) | 57.6 (22.6)
  30 Day change from Baseline SF-12 Physical Summary | 5.1 (10.5) | 6.0 (10.0) | 3.3 (10.5) | 4.3 (9.8)
  30 Day change from Baseline SF-12 Mental Health S | 3.4 (12.5) | 2.3 (12.6) | 1.8 (11.3) | 3.2 (10.6)
  30 Day change from Baseline KC Overall Summary | 20.9 (24.2) | 20.2 (24.0) | 17.4 (25.6) | 18.3 (23.1)
  30 Day change from Baseline KC Clinical Summary | 17.4 (23.9) | 16.6 (22.9) | 15.2 (24.5) | 14.8 (22.2)
  6M change from Baseline SF-12 Physical Summary | 5.8 (10.8) | 5.6 (10.1) | 3.6 (9.8) | 4.7 (10.7)
  6M change from Baseline SF-12 Mental Health Sum | 3.3 (11.2) | 3.3 (12.6) | 2.8 (10.5) | 3.3 (11.6)
  6M change from Baseline KC Overal Summary Score | 22.9 (23.8) | 22.7 (22.6) | 23.5 (25.5) | 21.2 (23.1)
  6M change from Baseline KC Clinical Summary Score | 17.8 (22.7) | 17.0 (22.2) | 17.5 (24.0) | 15.9 (22.2)
  1Y change from Baseline SF-12 Physical Summary | 4.7 (10.9) | 5.2 (10.1) | 3.0 (10.8) | 3.7 (10.6)
  1Y change from Baseline SF-12 Mental Health Sum | 3.5 (11.5) | 3.7 (12.9) | 3.2 (12.5) | 3.0 (11.1)
  1Y change from Baseline KC Overall Summary Score | 21.6 (24.4) | 21.4 (23.2) | 23.2 (26.7) | 20.0 (22.2)
  1Y change from Baseline KC Clinical Summary Score | 16.3 (23.8) | 15.0 (21.5) | 15.6 (26.8) | 14.0 (21.7)

15. Other Pre Specified Outcome: Percentage of Participants With Mortality
Description: All-cause, Cardiovascular, and Non-cardiovascular
Time Frame: as for outcome 10
Population: Intent to Treat patients with mortality or who were event free with sufficient follow-up for the applicable time point (30 days - at least 23 days of follow-up; 6 months - at least 150 days of follow-up; 1 year - at least 335 days of follow-up).
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge All Cause Mortality | 1.3 | 2.0 | 0.0 | 2.0
  Discharge Cardiovascular Mortality | 1.3 | 2.0 | 0.0 | 2.0
  Discharge Non-Cardiovascular Mortality | 0.0 | 0.0 | 0.0 | 0.0
  30 Day All Cause Mortality: number analyzed (Participants) | 601 | 303 | 102 | 295
  30 Day All Cause Mortality | 2.5 | 2.3 | 0.0 | 3.4
  30 Day Cardiovascular Mortality: number analyzed (Participants) | 601 | 303 | 102 | 295
  30 Day Cardiovascular Mortality | 2.3 | 2.3 | 0.0 | 3.4
  30 Day Non-Cardiovascular Mortality: number analyzed (Participants) | 601 | 303 | 102 | 295
  30 Day Non-Cardiovascular Mortality | 0.2 | 0.0 | 0.0 | 0.0
  6 Month All Cause Mortality: number analyzed (Participants) | 594 | 300 | 102 | 295
  6 Month All Cause Mortality | 7.7 | 8.3 | 8.8 | 7.1
  6 Month Cardiovascular Mortality: number analyzed (Participants) | 594 | 300 | 102 | 295
  6 Month Cardiovascular Mortality | 5.6 | 6.7 | 5.9 | 4.7
  6 Month Non-Cardiovascular Mortality: number analyzed (Participants) | 594 | 300 | 102 | 295
  6 Month Non-Cardiovascular Mortality | 2.2 | 1.7 | 2.9 | 2.4
  1 Year All Cause Mortality: number analyzed (Participants) | 587 | 297 | 101 | 293
  1 Year All Cause Mortality | 11.9 | 13.5 | 12.9 | 9.2
  1 Year Cardiovascular Mortality: number analyzed (Participants) | 587 | 297 | 101 | 293
  1 Year Cardiovascular Mortality | 7.7 | 9.8 | 7.9 | 5.8
  1 Year Non-Cardiovascular Mortality: number analyzed (Participants) | 587 | 297 | 101 | 293
  1 Year Non-Cardiovascular Mortality | 4.3 | 3.7 | 5.0 | 3.4

16. Other Pre Specified Outcome: Percentage of Participants With Stroke
Description: Disabling Stroke and Non-disabling Stroke
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge All Stroke | 4.4 | 4.3 | 3.9 | 5.4
  Discharge Disabling Stroke | 1.8 | 3.3 | 3.9 | 3.7
  Discharge Non-Disabling Stroke | 2.6 | 1.0 | 0.0 | 1.7
  30 Day All Stroke | 4.8 | 4.3 | 4.9 | 6.8
  30 Day Disabling Stroke | 2.0 | 3.3 | 3.9 | 4.4
  30 Day Non-Disabling Stroke | 2.8 | 1.0 | 1.0 | 2.4
  6 Month All Stroke | 5.9 | 8.3 | 6.9 | 8.1
  6 Month Disabling Stroke | 2.7 | 6.3 | 5.9 | 5.4
  6 Month Non-Disabling Stroke | 3.2 | 2.0 | 1.0 | 2.7
  1 Year All Stroke | 7.0 | 9.4 | 7.9 | 8.5
  1 Year Disabling Stroke | 3.6 | 7.1 | 5.9 | 5.8
  1 Year Non-Disabling Stroke | 3.6 | 2.4 | 2.0 | 2.7

17. Other Pre Specified Outcome: Percentage of Participants With Myocardial Infarction (MI)
Description: Periprocedural (≤72 hours post index procedure) and spontaneous (>72 hours post index procedure)
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge Myocardial Infarction | 0.5 | 1.6 | 2.0 | 0.7
  Discharge Peri-procedural MI | 0.5 | 1.3 | 2.0 | 0.7
  Discharge Spontaneous MI | 0.0 | 0.3 | 0.0 | 0.0
  30 Day Myocardial Infarction | 0.7 | 1.3 | 2.0 | 1.0
  30 Day Peri-procedural MI | 0.5 | 1.0 | 2.0 | 0.7
  30 Day Spontaneous MI | 0.2 | 0.3 | 0.0 | 0.3
  6 Month Myocardial Infarction | 2.0 | 3.0 | 2.9 | 3.7
  6 Month Peri-procedural MI | 0.5 | 1.3 | 2.0 | 0.7
  6 Month Spontaneous MI | 1.5 | 2.0 | 1.0 | 3.1
  1 Year Myocardial Infarction | 3.2 | 4.4 | 5.0 | 4.4
  1 Year Peri-procedural MI | 0.5 | 1.3 | 2.0 | 0.7
  1 Year Spontaneous MI | 2.7 | 3.4 | 3.0 | 3.8

18. Other Pre Specified Outcome: Percentage of Participants With Bleeding
Description: Life-threatening (or disabling) and major (defined below)
  Life-threatening or Disabling Bleeding
  * Fatal bleeding (Bleeding Academic Research Consortium [BARC] type 5124,125)
  * Bleeding in a critical organ, such as intracranial, intraspinal, intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome (BARC type 3b and 3c)
  * Bleeding causing hypovolemic shock or severe hypotension requiring vasopressors or surgery (BARC type 3b)
  * Overt source of bleeding with drop in hemoglobin of ≥5 g/dL or whole blood or packed red blood cells (RBC) transfusion ≥4 units (BARC type 3b)
  Major Bleeding (BARC type 3a)
  * Overt bleeding either associated with a drop in the hemoglobin level of at least 3.0g/dL or requiring transfusion of 2 or 3 units of whole blood/RBC, or causing hospitalization or permanent injury, or requiring surgery AND does not meet criteria of life-threatening or disabling bleeding
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge Bleeding | 11.9 | 10.5 | 8.8 | 9.5
  Discharge Life-threatening or Disabling Bleeding | 7.2 | 5.9 | 7.8 | 5.4
  Discharge Major Bleeding | 4.6 | 4.6 | 1.0 | 4.1
  30 Day Bleeding | 12.8 | 10.9 | 11.8 | 11.9
  30 Day Life-threatening or Disabling Bleeding | 8.0 | 5.0 | 9.8 | 6.1
  30 Day Major Bleeding | 4.8 | 5.9 | 2.0 | 5.8
  6 Month Bleeding | 16.5 | 17.0 | 17.6 | 14.9
  6 Month Life-threatening or Disabling Bleeding | 9.3 | 9.0 | 14.7 | 8.5
  6 Month Major Bleeding | 7.2 | 8.0 | 2.9 | 6.8
  1 Year Bleeding | 18.1 | 17.8 | 20.8 | 19.1
  1 Year Life-threatening or Disabling Bleeding | 9.9 | 9.8 | 16.8 | 11.3
  1 Year Major Bleeding | 8.3 | 8.4 | 5.0 | 8.9

19. Other Pre Specified Outcome: Percentage of Participants With Acute Kidney Injury
Description: Acute kidney injury based on the AKIN System Stage 3 (including renal replacement therapy) or Stage 2
  Change in serum creatinine (up to 7 days) compared to baseline:
  * Stage 1: Increase in serum creatinine to 150-199% (1.5-1.99 × increase compared with baseline) OR increase of ≥0.3 mg/dl (≥26.4 mmol/L)
  * Stage 2: Increase in serum creatinine to 200-299% (2.0-2.99 × increase compared with baseline)
  * Stage 3: Increase in serum creatinine to ≥300% (>3 × increase compared with baseline) OR serum creatinine of ≥4.0 mg/dL (≥354 mmol/L) with an acute increase of at least 0.5 mg/dL (44 mmol/L)
  -OR-
  Based on urine output (up to 7 days):
  * Stage 1: <0.5 ml/kg per hour for >6 but <12 hours
  * Stage 2: <0.5 ml/kg per hour for >12 but <24 hours
  * Stage 3: <0.3 ml/kg per hour for ≥24 hours or anuria for ≥12 hours
  Note 1: Subjects receiving renal replacement therapy are considered to meet Stage 3 criteria irrespective of other criteria.
Time Frame: ≤7 days post index procedure
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Acute Kidney Injury - Stage 2 or Stage 3 | 2.3 | 3.6 | 1.0 | 0.7
  Stage 2 | 1.0 | 1.3 | 0.0 | 0.0
  Stage 3 (including renal replacement therapy) | 1.3 | 2.3 | 1.0 | 0.7

20. Other Pre Specified Outcome: Percentage of Participants With Major Vascular Complication
Description: Major vascular complication - including access site related and non access site related
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge Major Vascular Complications | 6.8 | 5.6 | 8.8 | 7.8
  Discharge Access Site Related | 4.6 | 3.6 | 6.9 | 4.4
  Discharge Not Access Site Related | 2.3 | 2.0 | 2.9 | 3.4
  30 Day Major Vascular Complications | 7.0 | 5.3 | 8.8 | 7.8
  30 Day Access Site Related | 4.7 | 3.3 | 6.9 | 4.4
  30 Day Not Access Site Related | 2.5 | 2.0 | 2.9 | 3.4
  6 Month Major Vascular Complications | 7.6 | 5.7 | 8.8 | 8.1
  6 Month Access Site Related | 5.1 | 3.7 | 6.9 | 4.4
  6 Month Not Access Site Related | 2.7 | 2.0 | 2.9 | 3.7
  1 Year Major Vascular Complications | 7.7 | 6.1 | 8.9 | 8.2
  1 Year Access Site Related | 5.1 | 3.7 | 6.9 | 4.8
  1 Year Not Access Site Related | 2.7 | 2.4 | 3.0 | 3.8

21. Other Pre Specified Outcome: Percentage of Participants With Repeat Procedure for Valve-related Dysfunction
Description: Repeat procedure for valve-related dysfunction (surgical or interventional therapy)
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge Repeat proc valve-related dysfunction | 0.0 | 0.7 | 1.0 | 0.3
  30 Day Repeat proc valve-related dysfunction | 0.0 | 1.0 | 1.0 | 0.7
  6 Month Repeat proc valve-related dysfunction | 0.2 | 1.7 | 1.0 | 1.0
  1 Year Repeat proc valve-related dysfunction | 0.2 | 2.0 | 1.0 | 1.0

22. Other Pre Specified Outcome: Percentage of Participants With Hospitalization for Valve-related Symptoms or Worsening Congestive Heart Failure
Description: Hospitalization for valve-related symptoms or worsening congestive heart failure (New York Hear Association [NYHA] class III or IV)
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge | 0.8 | 0.7 | 1.0 | 0.0
  30 Day | 1.7 | 3.0 | 4.9 | 2.4
  6 Month | 6.7 | 9.3 | 9.8 | 6.4
  1 Year | 11.2 | 13.8 | 13.9 | 9.6

23. Other Pre Specified Outcome: Percentage of Participants With New Permanent Pacemaker Implantation
Description: New permanent pacemaker implantation resulting from new or worsened conduction disturbances
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge | 28.2 | 14.8 | 27.5 | 24.1
  30 Day | 29.1 | 15.8 | 28.4 | 28.1
  6 Month | 33.3 | 18.0 | 29.4 | 30.2
  1 Year | 34.2 | 18.5 | 30.7 | 31.1

24. Other Pre Specified Outcome: Percentage of Participants With New Onset of Atrial Fibrillation or Atrial Flutter
Description: New onset of atrial fibrillation or atrial flutter
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge | 6.4 | 3.9 | 4.9 | 5.1
  30 Day | 5.8 | 4.3 | 5.9 | 5.1
  6 Month | 6.6 | 4.7 | 5.9 | 5.1
  1 Year | 6.6 | 4.7 | 5.9 | 5.1

25. Other Pre Specified Outcome: Percentage of Participants With Coronary Obstruction
Description: Coronary obstruction
Time Frame: ≤72 hours post index procedure
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants | 0.2 | 0.7 | 1.0 | 0.7

26. Other Pre Specified Outcome: Percentage of Participants With Ventricular Septal Perforation
Description: Ventricular septal perforation
Time Frame: ≤72 hours post index procedure
Population: Intent to Treat
Measure: Number; unit: Percentage of participant
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participant | 0.2 | 0.0 | 0.0 | 0.0

27. Other Pre Specified Outcome: Percentage of Participants With Mitral Apparatus Damage
Description: Mitral apparatus damage
Time Frame: ≤72 hours post index procedure
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants | 0.0 | 0.3 | 0.0 | 0.0

28. Other Pre Specified Outcome: Percentage of Participants With Cardiac Tamponade
Description: Cardiac tamponade
Time Frame: ≤72 hours post index procedure
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants | 2.5 | 1.3 | 2.0 | 1.4

29. Other Pre Specified Outcome: Percentage of Participants With Prosthetic Aortic Valve Malpositioning
Description: Prosthetic aortic valve malpositioning, including valve migration, valve embolization, or ectopic valve deployment
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge Prosthetic aortic valve malpositioning | 0.0 | 2.6 | 0.0 | 0.0
  Discharge Valve Migration | 0.0 | 0.7 | 0.0 | 0.0
  Discharge Valve Embolization | 0.0 | 2.0 | 0.0 | 0.0
  Discharge Ectopic Valve Deployment (Procedural) | 0.0 | 0.3 | 0.0 | 0.0
  30 Day Prosthetic aortic valve malpositioning | 0.0 | 2.6 | 0.0 | 0.0
  30 Day Valve Migration | 0.0 | 0.7 | 0.0 | 0.0
  30 Day Valve Embolization | 0.0 | 2.0 | 0.0 | 0.0
  30 Day Ectopic Valve Deployment (Procedural) | 0.0 | 0.3 | 0.0 | 0.0
  6 Month Prosthetic aortic valve malpositioning | 0.0 | 2.7 | 0.0 | 0.0
  6 Month Valve Migration | 0.0 | 0.7 | 0.0 | 0.0
  6 Month Valve Embolization | 0.0 | 2.0 | 0.0 | 0.0
  6 Month Ectopic Valve Deployment (Procedural) | 0.0 | 0.3 | 0.0 | 0.0
  1 Year Prosthetic aortic valve malpositioning | 0.0 | 2.7 | 0.0 | 0.0
  1 Year Valve Migration | 0.0 | 0.7 | 0.0 | 0.0
  1 Year Valve Embolization | 0.0 | 2.0 | 0.0 | 0.0
  1 Year Ectopic Valve Deployment (Procedural) | 0.0 | 0.3 | 0.0 | 0.0

30. Other Pre Specified Outcome: Percentage of Participants With Prosthetic Aortic Valve Thrombosis
Description: Prosthetic aortic valve thrombosis
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge | 0.0 | 0.0 | 0.0 | 1.0
  30 Day | 0.0 | 0.0 | 1.0 | 1.4
  6 Month | 1.2 | 0.0 | 3.9 | 2.0
  1 Year | 1.5 | 0.0 | 6.9 | 2.4

31. Other Pre Specified Outcome: Percentage of Participants With Prosthetic Aortic Valve Endocarditis
Description: Prosthetic aortic valve endocarditis
Time Frame: as for outcome 10
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
Number analyzed (Participants) | 607 | 305 | 102 | 295
Percentage of participants
  Discharge | 0.0 | 0.0 | 0.0 | 0.0
  30 Day | 0.2 | 0.0 | 0.0 | 0.0
  6 Month | 0.5 | 0.0 | 3.9 | 0.3
  1 Year | 0.7 | 0.0 | 4.0 | 0.3

ADVERSE EVENTS:
Time Frame: 1 Year
Description: For All Cause Mortality, the at risk population (denominator) is the ITT population who had the event or who were event free with sufficient follow-up (at least 335 days of follow-up).
  For the SAE/AE tables, the at risk population (denominator) is the full ITT population.
Arm/Group | Lotus Valve System - Randomized | CoreValve TAVR System - Randomized | Lotus Valve System - Single-arm Roll-in Cohort | Lotus Valve System - Single-arm Continued Access Cohort
All-Cause Mortality (participants affected / at risk) | 70/587 | 40/297 | 13/101 | 27/293
Serious Adverse Events (participants affected / at risk) | 431/607 | 207/305 | 72/102 | 229/295
Other Adverse Events (participants affected / at risk) | 458/607 | 210/305 | 83/102 | 228/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotus Valve System - Randomized (N=607) | CoreValve TAVR System - Randomized (N=305) | Lotus Valve System - Single-arm Roll-in Cohort (N=102) | Lotus Valve System - Single-arm Continued Access Cohort (N=295)
Anaemia (Blood and lymphatic system disorders) | 27 (27) | 5 (5) | 4 (4) | 8 (8)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 8 (8) | 9 (9) | 0 (0) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 3 (3) | 9 (9)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 135 (135) | 37 (37) | 19 (19) | 62 (62)
Cardiac failure congestive (Cardiac disorders) | 62 (75) | 38 (54) | 11 (14) | 23 (24)
Atrial fibrillation (Cardiac disorders) | 28 (28) | 7 (7) | 6 (6) | 17 (20)
Bundle branch block left (Cardiac disorders) | 22 (22) | 9 (9) | 8 (8) | 15 (15)
Cardiac arrest (Cardiac disorders) | 16 (16) | 4 (4) | 3 (4) | 7 (8)
Cardiac failure (Cardiac disorders) | 13 (15) | 7 (7) | 1 (1) | 4 (4)
Atrioventricular block (Cardiac disorders) | 14 (14) | 9 (9) | 7 (7) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 12 (13) | 8 (8) | 0 (0) | 11 (11)
Conduction disorder (Cardiac disorders) | 12 (12) | 8 (8) | 1 (1) | 5 (5)
Bradycardia (Cardiac disorders) | 9 (9) | 3 (3) | 1 (1) | 7 (7)
Pericardial effusion (Cardiac disorders) | 9 (9) | 5 (5) | 1 (1) | 4 (4)
Atrioventricular block second degree (Cardiac disorders) | 8 (8) | 3 (3) | 0 (0) | 7 (7)
Sick sinus syndrome (Cardiac disorders) | 8 (8) | 3 (3) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 6 (6) | 8 (8) | 1 (1) | 4 (4)
Cardiac tamponade (Cardiac disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 3 (5) | 3 (4) | 1 (1) | 4 (4)
Atrioventricular block first degree (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 4 (4) | 3 (3) | 3 (3) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Mitral valve incompetence (Cardiac disorders) | 2 (3) | 1 (1) | 2 (3) | 1 (1)
Angina unstable (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Mitral perforation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electromechanical dissociation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial rupture (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve calcification (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trifascicular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular asystole (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peutz-Jeghers syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (12) | 9 (9) | 5 (5) | 10 (11)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 4 (4) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 3 (3)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 8 (8) | 3 (3) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 7 (7) | 4 (4) | 0 (0) | 3 (3)
Asthenia (General disorders) | 5 (5) | 1 (1) | 4 (4) | 3 (3)
Adverse drug reaction (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Catheter site necrosis (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 2 (2) | 1 (1) | 2 (2) | 8 (8)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Implant site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hernia obstructive (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical complication of implant (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 23 (25) | 13 (14) | 4 (4) | 15 (16)
Sepsis (Infections and infestations) | 18 (18) | 5 (5) | 1 (1) | 7 (7)
Urinary tract infection (Infections and infestations) | 10 (10) | 9 (9) | 4 (5) | 9 (11)
Septic shock (Infections and infestations) | 6 (6) | 4 (4) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 5 (5) | 2 (2) | 4 (4) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 3 (4) | 1 (1) | 3 (3) | 2 (2)
Catheter site infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Staphylococcal sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Catheter site cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected sebaceous cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 26 (26) | 16 (16) | 3 (4) | 14 (14)
Vascular access complication (Injury, poisoning and procedural complications) | 12 (12) | 4 (4) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 5 (5) | 0 (0) | 5 (5)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 6 (6) | 3 (3) | 1 (1) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 2 (2) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 1 (1) | 3 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lead dislodgement (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pacemaker complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Frostbite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Post procedural stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device lead damage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Echocardiogram abnormal (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine cytology abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood culture positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus rhythm (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulse absent (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile toxin test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pedal pulse decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 1 (1) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 21 (21) | 20 (20) | 5 (5) | 14 (14)
Syncope (Nervous system disorders) | 13 (13) | 7 (9) | 1 (1) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 8 (8) | 4 (4) | 1 (2) | 6 (6)
Embolic stroke (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 3 (3) | 4 (5) | 1 (1) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 5 (5)
Dementia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chorea (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain stem syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polydipsia psychogenic (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 32 (33) | 15 (15) | 5 (5) | 9 (10)
Renal failure (Renal and urinary disorders) | 6 (6) | 4 (4) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (5) | 5 (6) | 5 (6) | 4 (6)
Urinary retention (Renal and urinary disorders) | 3 (3) | 4 (4) | 4 (4) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 7 (7) | 1 (1) | 10 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (5) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (5) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 13 (13) | 3 (3) | 9 (9)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2) | 0 (0) | 4 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 1 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 4 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 1 (1) | 4 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 2 (2) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activities of daily living impaired (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 8 (8) | 1 (1) | 0 (0) | 5 (5)
Hypertensive crisis (Vascular disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4) | 2 (3) | 1 (2) | 1 (2)
Intermittent claudication (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2) | 1 (1) | 5 (6)
Shock haemorrhagic (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Labile blood pressure (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iliac artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extravasation blood (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic macroangiopathy (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotus Valve System - Randomized (N=607) | CoreValve TAVR System - Randomized (N=305) | Lotus Valve System - Single-arm Roll-in Cohort (N=102) | Lotus Valve System - Single-arm Continued Access Cohort (N=295)
Thrombocytopenia (Blood and lymphatic system disorders) | 146 (149) | 42 (43) | 26 (26) | 67 (69)
Anaemia (Blood and lymphatic system disorders) | 86 (88) | 50 (56) | 13 (14) | 49 (51)
Leukocytosis (Blood and lymphatic system disorders) | 37 (38) | 25 (26) | 0 (0) | 17 (17)
Bundle branch block left (Cardiac disorders) | 227 (229) | 83 (87) | 40 (40) | 102 (103)
Atrial fibrillation (Cardiac disorders) | 58 (61) | 29 (30) | 11 (12) | 33 (33)
Cardiac failure congestive (Cardiac disorders) | 46 (53) | 18 (18) | 12 (13) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 44 (44) | 24 (24) | 6 (7) | 34 (35)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 16 (16)
Catheter site haematoma (General disorders) | 38 (38) | 22 (24) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 29 (30) | 18 (20) | 0 (0) | 22 (24)
Catheter site haemorrhage (General disorders) | 27 (29) | 21 (22) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 62 (66) | 34 (37) | 15 (16) | 28 (32)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 30 (31) | 17 (18) | 11 (11) | 20 (21)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Echocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 18 (18)
Hypervolaemia (Metabolism and nutrition disorders) | 35 (35) | 19 (19) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 29 (31) | 17 (19) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 27 (29) | 18 (19) | 0 (0) | 21 (23)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6) | 26 (28)
Renal failure acute (Renal and urinary disorders) | 55 (64) | 32 (42) | 0 (0) | 32 (33)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 41 (41) | 18 (18) | 6 (6) | 19 (19)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (16)
Hypertension (Vascular disorders) | 61 (65) | 37 (37) | 0 (0) | 29 (29)
Hypotension (Vascular disorders) | 56 (57) | 19 (20) | 13 (13) | 37 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT02202434/Prot_SAP_000.pdf